CLINICAL TRIAL: NCT06866197
Title: A Multi-Cohort, Prospective Investigation of the Symani® Surgical System: A Novel Approach to the Next Frontier of Microsurgery and Expanding Access to Care in Free Tissue Transfer and Lymphatic Surgery
Brief Title: CONNECT: A Multi-Cohort, Prospective Investigation of the Symani® Surgical System
Acronym: CONNECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDC-00145
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Microsurgery; Lymphedema; Free Tissue Transfer
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free Tissue Transfer, Therapeutic Lymphatic Surgery, Prophylactic Lymphatic Surgery Participants (Experimental)
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — The Symani Surgical System (Symani) is designed for open microsurgery procedures, featuring articulated and interchangeable instruments.

SUMMARY:
The objective of this clinical study is to evaluate the Symani System's safety and effectiveness for microsurgical anastomosis during free tissue transfer surgery and lymphatic surgery.

The primary endpoints are:

Effectiveness: Clinical Success, defined as intraoperative anastomosis patency. Safety: Freedom from device-related serious adverse events prior to discharge from the index hospitalization, as adjudicated by a Clinical Events Committee.

Participants will receive treatment as standard of care and be asked to:

Allow the researchers to access and use their information. If participants are undergoing a therapeutic lymphatic procedure, they will be asked to complete a questionnaire and undergo lymphedema volume assessments as part of the study. If participants are undergoing a prophylactic lymphatic procedure, they will only be asked to undergo limb volume assessments.

Participants will be asked to comply with the follow-up visits as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults, according to the local law
* Patient agrees to participate in the study, return for all required follow-up visits, and has willingly provided written informed consent after receiving all information related to the study, its requirements, and the robotic assisted procedure
* Patient with a clinical indication for a microsurgical anastomosis for a free flap transfer surgery and/or lymphatic surgery Investigator considers candidate acceptable for free flap transfer surgery and/or lymphatic surgery with a robotic assisted microsurgical anastomosis in accordance with the Symani System IFU

Inclusion Criteria for Therapeutic Lymphatic Patients:

* For lymphedema of the extremities, swelling of lymphedema that is not completely reversed by decongestion therapy modalities. (Not applicable for patients with lymphedema of the head and neck)
* For lymphedema of the extremities, at least one of the following positive quantitative measurements (not applicable for patients with lymphedema of the head and neck):

  1. Volumetry differential between diseased limb and contralateral limb must be at least 10% of the other
  2. Bioimpedance (L-Dex) differential, if feasible, between diseased limb and contralateral limb of at least 10 units
* Maintain complete decongestive therapy (CDT), according to International Society of Lymphology (ISL) guidelines, for a minimum duration of four (4) weeks prior to screening
* Willingness to comply with recommended regimen of self-care, with consistent use of compression garments from screening through the entire study duration
* Patient must be diagnosed with Lymphedema
* Patient must have a body mass index (BMI) of ≤ 35

Inclusion Criteria for Prophylactic Lymphatic Patients:

* The patient has at least one identifiable risk factor for developing lymphedema of the extremities
* Patient with a body mass index (BMI) of ≤ 35

Exclusion Criteria:

* Patients who are not capable and/or unwilling to provide informed consent
* Clinically significant cardiovascular, digestive, respiratory, endocrine, liver or central nervous system disorders, previous mental disorders, or other disorders that may significantly affect the data collection or the ability to comply with the protocol per the investigators discretion.
* Known history of significant bleeding, coagulopathy, or Von Willebrand's disease
* Patients with implanted pacemaker
* Planned vein graft (either venous or arterial)
* Previously documented history of chronic kidney disease (eGFR ≤ 30)
* Currently enrolled in any other investigational clinical studies that the investigator believes may impact patient safety or outcomes
* Patients belonging to vulnerable populations, such as pregnant women, or patients ineligible to participate for other reasons in the judgement of the investigator

Exclusion Criteria for Free Tissue Transfer Patients:

* Patients with buried flaps
* Multiple flaps planned for the procedure

Exclusion Criteria for Therapeutic Lymphatic Patients:

* Patients with venous edema (arising from increased capillary filtration)
* Patients with other medical conditions that could lead to acute limb edema, such as (but not limited to) acute venous thrombosis or heart failure
* Current infection in the affected area of lymphedema
* Current evidence of malignancy
* Known iodine sensitivity
* Patient's lymphatic disease is due to lipedema
* Patients with bilateral lymphedema or lymphedema in multiple anatomical locations

Exclusion Criteria for Prophylactic Lymphatic Participants:

* Patients for whom prophylactic surgery on more than one limb is planned
* Known iodine sensitivity
* Patients with post-thrombotic syndrome, arterial insufficiency, deep vein thrombosis or any other medical condition that could make them ineligible to participate in the judgment of the investigator
* Patients diagnosed with lymphedema

Intraoperative Exclusion Criteria:

* Any presenting condition discovered intraoperatively that, in the opinion of the investigator, would make participating in this study not in the patient's best interest
* The patient does not have at least two robotic sutures attempted during the index procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2028-02-03 (Estimated); Study Completion 2029-02-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Success, defined as intraoperative anastomosis patency. | The duration of the participants' index procedure, from when they enter the OR to when they leave the OR (procedures typically last under 24 hours)
  Clinical Success is defined as intraoperative anastomosis patency. Intraoperative anastomosis patency will be measured for each robotic anastomosis per standard of care and will be evaluated prior to closure of the procedure site during the index procedure.
Freedom from device-related serious adverse events prior to discharge from the index hospitalization | The duration of the participants' index procedure hospitalization (typically lasting under two weeks)
  Freedom from device-related serious adverse events prior to discharge from the index hospitalization. All device-related serious adverse events will be descriptively summarized.

SECONDARY OUTCOMES:
Freedom from a reoperation to revise a robotic anastomosis prior to discharge | The duration of the participants' index procedure hospitalization (typically lasting under two weeks)
  Freedom from returning to the operating room for surgical revisions to an anastomosis that was deemed robotic in the index procedure. This endpoint will be evaluated at discharge for each participant.
Rate of intra-operative approach changes from robotic to manual | The duration of the participants' index procedure, from when they enter the OR to when they leave the OR (procedures typically last under 24 hours).
  An intra-operative approach change is defined as a conversion from a robotic anastomosis approach to a manual anastomosis approach. This endpoint will be evaluated upon completion of the index procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Vincent's Hospital Melbourne, Melbourne, Victoria, Australia